CLINICAL TRIAL: NCT02321839
Title: Evaluation of the Usefulness of a Treat and Extend Regimen Using Ranibizumab for Neovascular Age-Related Macular Degeneration.
Brief Title: Evaluation of the Usefulness of a Treat and Extend Regimen Using Ranibizumab for Neovascular AMD.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nagoya City University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Yuichiro Ogura, Professor, Nagoya City University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAENCU001
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2016-10

CONDITIONS: Neovascular Age-related Macular Degeneration
Keywords: neovascular age-related macular degeneration; Ranibizumab; Treat and extend

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intraviteal Ranibizumab 0.5mg (Experimental): Intraviteal Ranibizumab 0.5mg
  Interventions: Drug: Intraviteal Ranibizumab 0.5mg

INTERVENTIONS:
Drug: Intraviteal Ranibizumab 0.5mg — Intraviteal Ranibizumab 0.5mg

SUMMARY:
To evaluate the visual outcome, number of injections and visits, and the effect of mental status of a treat and extend regimen in managing neovascular age-related macular degeneration with intravitreal ranibizumab.

DETAILED DESCRIPTION:
Treat and Extend Regimen (TER) may contribute to the improvement to a patients' mentality, since the treatment intervals are extended if there were no signs of recurrence. Therefore, we have planned to examine the psychological impact of TER using Hospital Anxiety and Depression Scale (HADS), in addition to the improvement of visual acuity and central retinal thickness.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Male or female of aged 50 years or older
* Typical AMD and PCV patients
* BCVA of 24 letters or over

Exclusion Criteria:

* Total lesion area of >12 DA or >30.5 mm2
* The existence of subretinal hemorrhage area constituting ≥50% of total lesion area
* The existence of scar or fibrosis area constituting ≥50% of total lesion area
* The existence of RPE tear
* Prior treatment for wet AMD
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD
* The pregnant or lactating woman

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-01; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Visual acuity | One Year

SECONDARY OUTCOMES:
central foveal thickness | One and two years

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale | one and two years
  The mean change from baseline in Hospital Anxiety and Depression Scale at week 52 and 104.

CONTACTS AND LOCATIONS:
Overall Officials: Yuichiro Ogura, Study Chair — Nagoya City Univsersity
Locations (2):
- Japan (2):
  - Sugita Eye Hospital, Nagoya, Aichi-ken
  - Nagoya City Univsersity, Nagoya, Aichi-ken

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kato A, Yasukawa T, Sugita I, Yoshida M, Nozaki M, Hirano Y, Kondo J, Abe T, Sugita K, Okita T, Morita H, Takase N, Ogura Y. Mental Status and Feasibility of an Intravitreal Ranibizumab Treat-and-Extend Regimen in Patients with Neovascular Age-Related Macular Degeneration. Adv Ther. 2022 Mar;39(3):1403-1416. doi: 10.1007/s12325-022-02052-1. Epub 2022 Feb 3. PMID 35112307